CLINICAL TRIAL: NCT06788600
Title: An EBV mRNA Vaccine (WGc-043 Injection) in Patients With EB Virus-positive Relapsed or Refractory Lymphoma: A Phase I Clinical Trial Assessing the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Preliminary Anti-tumor Activity
Brief Title: Mechanistic Study of EBV mRNA Vaccine (WGc-043) in EBV-Positive Relapsed/Refractory Lymphoma
Acronym: WGc-043
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, MD, Ruijin Hospital
Other Study IDs: mRNAvaccine-WGc-043
Record Dates: First submitted 2025-01-13; First posted 2025-01-23 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-01

CONDITIONS: Epstein-Barr Virus Associated Lymphoma
Keywords: relapsed or refractory lymphoma; Epstein-Barr virus mRNA vaccine; Epstein-Barr virus-positive lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- EBV mRNA vaccine infusion with a dose of 100 µg: Drug: EBV mRNA vaccine (WGc-043) Patients will receive a 100 µg dose of the EBV mRNA vaccine per administration, including 5 doses for the primary immunization regimen and subsequent optional personalized treatment. For the primary immunization, the first 4 doses will be administered weekly, with the 5th dose given 4 weeks after the 4th dose.
  Interventions: Drug: EBV mRNA vaccine (WGc-043)
- EBV mRNA vaccine infusion with a dose of 200 µg: Drug: EBV mRNA vaccine (WGc-043) Patients will receive a 200 µg dose of the EBV mRNA vaccine per administration, including 5 doses for the primary immunization regimen and subsequent optional personalized treatment. For the primary immunization, the first 4 doses will be administered weekly, with the 5th dose given 4 weeks after the 4th dose.
  Interventions: Drug: EBV mRNA vaccine (WGc-043)
- EBV mRNA vaccine infusion with a dose of 300 µg: Drug: EBV mRNA vaccine (WGc-043) Patients will receive a 300 µg dose of the EBV mRNA vaccine per administration, including 5 doses for the primary immunization regimen and subsequent optional personalized treatment. For the primary immunization, the first 4 doses will be administered weekly, with the 5th dose given 4 weeks after the 4th dose.
  Interventions: Drug: EBV mRNA vaccine (WGc-043)
- EBV mRNA vaccine infusion with a dose of 400 µg: Drug: EBV mRNA vaccine (WGc-043) Patients will receive a 400 µg dose of the EBV mRNA vaccine per administration, including 5 doses for the primary immunization regimen and subsequent optional personalized treatment. For the primary immunization, the first 4 doses will be administered weekly, with the 5th dose given 4 weeks after the 4th dose.
  Interventions: Drug: EBV mRNA vaccine (WGc-043)

INTERVENTIONS:
Drug: EBV mRNA vaccine (WGc-043) — Each subject will be infused with EBV mRNA vaccine per administration, including 5 doses for the primary immunization regimen and subsequent optional personalized treatment. For the primary immunization, the first 4 doses will be administered weekly, with the 5th dose given 4 weeks after the 4th dose.
  The specific dose of mRNA vaccine will be determined according to the experimental group.

SUMMARY:
This exploratory study, based on a pharmaceutical company-initiated clinical trial, aims to investigate the therapeutic effects of the EBV mRNA vaccine (WGc-043 injection) in treating EBV-positive relapsed or refractory lymphoma. The study explores the mechanism of the EBV mRNA vaccine (WGc-043 injection) within the tumor microenvironment in EBV-positive lymphoma, elucidating the vaccine's inhibitory effects on EBV. This research will provide a theoretical foundation for the application of mRNA vaccines, either alone or in combination with other immunotherapies, in the treatment of EBV-positive lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 75 years (inclusive).
2. Histologically or cytologically diagnosed as relapsed or refractory EBV-positive lymphoma (confirmed by in situ hybridization (ISH) or fluorescence in situ hybridization (FISH) showing EBER positivity in tumor tissue) that has failed standard treatment and lacks effective treatment options. This includes, but is not limited to, NK/T-cell lymphoma, Diffuse Large B-cell Lymphoma (DLBCL), or other Peripheral T-cell Lymphomas (PTCL).Relapse is defined as the appearance of new lesions in the primary site or elsewhere after achieving complete remission (CR).

(1)Refractory is defined by any of the following conditions: No partial response (PR) after ≥2 cycles of treatment. No CR after ≥4 cycles of treatment. No complete remission (CR) after autologous hematopoietic stem cell transplantation.

If the best response or reason for discontinuation is progressive disease (PD), no cycle number requirements apply.

(2)Prior treatment must include:

1. Relapsed/Refractory DLBCL: Must have received at least second-line systemic therapy.
2. Relapsed/Refractory Peripheral T-cell Lymphoma: Must have received at least first-line systemic therapy.
3. Relapsed/Refractory NK/T-cell Lymphoma: Must have received a regimen based on L-asparaginase (I/II stage diseases as per the nasal NK/T-cell lymphoma CA staging system must have also received radiotherapy).

   3.Eastern Cooperative Oncology Group (ECOG) Performance Status: 0-2 points. 4.Expected survival ≥3 months. 5.At least one measurable lesion as defined by the Lymphoma Classification (2014 version), with measurable lesions defined as:
   1. A lymph node lesion with a maximum long diameter >15 mm on enhanced CT, MRI, or PET-CT.
   2. An extranodal lesion with a maximum long diameter >10 mm. 6.Adequate organ function as evidenced by the following criteria:

   <!-- -->

   1. No use of granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), recombinant human erythropoietin, recombinant human thrombopoietin, or blood component transfusion within 14 days prior to screening. Hemoglobin ≥80 g/L; neutrophil count >1.0 × 10^9/L; platelet count ≥75 × 10^9/L.
   2. Total bilirubin ≤1.5× upper limit of normal (ULN); if liver metastasis or Gilbert's syndrome present, total bilirubin ≤3× ULN.
   3. ALT or AST ≤2.5× ULN; if liver metastasis, ALT or AST ≤5× ULN.
   4. Serum creatinine (SCr) ≤1.5× ULN or creatinine clearance ≥50 mL/min (Cockcroft-Gault formula).
   5. Prothrombin time (PT), International Normalized Ratio (INR) ≤1.5× ULN (unless using warfarin for anticoagulation).
   6. Cardiac Doppler ultrasound evaluation: Left ventricular ejection fraction (LVEF) ≥50%.
   7. If the investigator considers any of the above parameters below the study's lower limit due to disease progression, the patient's inclusion can be discussed with the sponsor and the CRO's medical team.

   7.No plans for pregnancy during the treatment period. Female patients of childbearing potential must have a negative pregnancy test and agree to use effective contraception during the trial and for 4 months after treatment.

   8.Able to understand and voluntarily sign a written informed consent form before the trial.

   9.Able to communicate well with the investigator and adhere to the protocol for completing the trial.

   Exclusion Criteria:

   - **Exclusion Criteria**
   1. Patients with a history of other tumors, except for skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, in situ cervical cancer, gastrointestinal mucosal carcinoma, or other malignancies considered acceptable by the investigator, provided these were treated and have not recurred within the last 5 years.
   2. Known to have aggressive NK-cell leukemia; central nervous system (CNS) lymphoma or CNS metastases; or associated hemophagocytic syndrome.
   3. Known to have poorly controlled cardiac clinical symptoms or diseases, such as NYHA Class II heart failure or higher (see Appendix 4, section 16.4), unstable angina, myocardial infarction within the past 6 months, or clinically significant and treatable supraventricular or ventricular arrhythmias.
   4. Any active autoimmune disease or history of autoimmune diseases, including but not limited to immune-related neurological diseases, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barré syndrome, myasthenia gravis, systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel diseases including Crohn's disease and ulcerative colitis, autoimmune hepatitis, toxic epidermal necrolysis (TEN), or Stevens-Johnson syndrome (except for Type 1 diabetes managed with stable doses of insulin).
   5. Any uncontrolled clinical disease (e.g., respiratory, circulatory, digestive, neurological, hematological, urogenital, endocrine diseases) or mental illness (e.g., depression, schizophrenia) or other significant illnesses that, in the investigator's assessment, could hinder informed consent, interfere with the interpretation of trial results, pose risks to the subject from participation, or otherwise affect the trial's objectives.
   6. History of interstitial lung disease or suspected interstitial lung disease; or presence of pulmonary abnormalities that may interfere with the detection or management of potential drug-related pulmonary toxicity during the trial.
   7. Allergies to the investigational drug (including any excipients). A history of severe allergic reactions to any drugs, foods, or vaccines, such as anaphylactic shock, allergic laryngeal edema, allergic dyspnea, allergic purpura, thrombocytopenic purpura, or local allergic necrotizing reactions (Arthus reactions).
   8. Any abnormalities at the injection site or permanent body art (e.g., tattoos) that the investigator believes may hinder observation of local reactions at the injection site.
   9. Contraindications to intramuscular injection (see Appendix 5, section 16.5).
   10. Less than 4 weeks since the last anti-tumor treatment (radiotherapy, chemotherapy, targeted therapy, immunotherapy, or local-regional therapy) or less than 2 weeks since palliative radiotherapy; patients with treatment-related adverse reactions (excluding hair loss) from previous anti-tumor therapy that have not recovered to NCI CTCAE ≤ 1 level.
   11. Previous organ transplantation or allogeneic hematopoietic stem cell transplantation.
   12. Systemic treatment with corticosteroids (>10 mg/day of prednisone or equivalent dose of other glucocorticoids) or other immunosuppressants within 14 days prior to the first dose of vaccine. However, inhaled or local use of steroids and adrenal hormone replacement at doses ≤10 mg/day of prednisone in the absence of active autoimmune disease is permitted.
   13. Receipt of an mRNA vaccine or similar nanoparticle delivery drugs (e.g., LNP) within 6 months prior to the first dose of vaccine.
   14. Receipt of live vaccines, attenuated live vaccines, or inactivated vaccines within 4 weeks prior to the first dose of vaccine.
   15. Previous administration of therapeutic vaccines or cellular immunotherapy for anti-tumor treatment.
   16. Participation in other clinical trials of drugs or devices within 3 months prior to screening.
   17. Blood donation or significant blood loss (>450 mL) within 3 months prior to screening.
   18. Major surgery within 4 weeks prior to screening (catheter placement or small biopsies as required by the protocol are not exclusion criteria), or if the impact of surgery or trauma has not resolved within 14 days prior to enrollment.
   19. History of substance abuse or known medical, psychological, or social conditions, such as a history of alcohol or drug abuse.
   20. Known infections with hepatitis B virus, hepatitis C virus, human immunodeficiency virus (HIV), or syphilis, or positive screening for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVAb), HIV antibody, or treponemal antibody (TP) at screening:

       * HBsAg(+) or HBcAb(+), with HBV DNA copy number ≥2000 IU/mL (or above the lower limit of positive detection at the study center);
       * HCVAb positive, with HCV RNA ≥ ULN at the study center.
   21. Patients with active tuberculosis (TB) (those suspected of having active TB must undergo chest X-ray, sputum tests, and exclude active TB through clinical symptoms and signs) or a history of active TB; or severe acute or chronic infections requiring systemic treatment.
   22. Pregnant or breastfeeding women.
   23. Any other factors that the investigator believes make the subject unsuitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with EBV-positive relapsed or refractory lymphoma
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
ScRNA-seq profiles of tumor tissues before and after injection | If the patient receives personalized treatment, safety follow-up will be conducted 28 days after the last infusion; if not, safety follow-up will be conducted 28 days after the 5th dose.
  Analysis of changes in the TME during treatment by comparing scRNA-seq profiles of tumor tissues before and after injection.
Clinical data from patients with disease remission (CR/PR) and those without remission (SD/PD) | If the patient receives personalized treatment, safety follow-up will be conducted 28 days after the last infusion; if not, safety follow-up will be conducted 28 days after the 5th dose.
  Identification of key molecular mechanisms and immune cell components associated with treatment efficacy by comparing data from patients with disease remission (CR/PR) and those without remission (SD/PD).

SECONDARY OUTCOMES:
Proportions of different immune cell types in tumor tissues from subjects with varying disease remission statuses. | If the patient receives personalized treatment, safety follow-up will be conducted 28 days after the last infusion; if not, safety follow-up will be conducted 28 days after the 5th dose.
  (1) Identification of immune cells associated with the formation of immune memory by comparing the proportions of different immune cell types in tumor tissues from subjects with varying disease remission statuses. The molecular mechanisms underlying this process will be explored through gene expression profiling, focusing on key immune cell components and molecular pathways related to T cell memory formation.
Gene expression profiling in tumor tissues from subjects with varying disease | If the patient receives personalized treatment, safety follow-up will be conducted 28 days after the last infusion; if not, safety follow-up will be conducted 28 days after the 5th dose.
  The molecular mechanisms underlying this process will be explored through gene expression profiling, focusing on key immune cell components and molecular pathways related to T cell memory formation. Identification of endogenous tumor factors associated with immune chemotaxis, T cell activation, and immune escape through correlation analysis with tumor cell characteristics, molecular genetic alterations, and oncogenic pathways.
Molecular biological changes in EBV in peripheral blood samples before and after EBV mRNA vaccine injection | Time Frame: If the patient receives personalized treatment, safety follow-up will be conducted 28 days after the last infusion; if not, safety follow-up will be conducted 28 days after the 5th dose.
  Analysis of molecular biological changes in EBV in peripheral blood samples before and after EBV mRNA vaccine injection, focusing on changes in genes, proteins, and other molecular markers.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No